CLINICAL TRIAL: NCT06119685
Title: Phase 1/2 Study of IDP-023 as a Single Agent and in Combination With Antibody Therapies in Patients With Advanced Hematologic Cancers
Brief Title: IDP-023 as a Single Agent and in Combination With Antibody Therapies in Patients With Advanced Hematologic Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indapta Therapeutics, INC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Indapta-Trial-1
Record Dates: First submitted 2023-10-22; First posted 2023-11-07 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-08

CONDITIONS: NHL; Multiple Myeloma; Blood Cancer; Refractory Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Multiple Myeloma; Relapsed Multiple Myeloma
Keywords: Advanced Hematologic Cancers
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms; Lymphoma, Non-Hodgkin | interventions — Rituximab; daratumumab; Interleukin-2; aldesleukin; Cyclophosphamide; fludarabine; Mesna; isatuximab

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose, and dose-expansion study of IDP-023 administered as a single agent and in combination with or without interleukin-2 (IL-2), and with or without isatuximab, daratumumab or rituximab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1: Single Agent IDP-023 - Single Dose (Experimental): NHL or MM patient treated with a single dose of IDP-023 monotherapy
  Interventions: Drug: IDP-023; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase 1: Single Agent IDP-023 - Multiple Doses (Experimental): NHL and MM patients treated with multiple doses of IDP-023 monotherapy
  Interventions: Drug: IDP-023; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase 1: Single Agent IDP-023 - Multiple Doses with IL-2 (Experimental): NHL and MM patients treated with multiple doses of IDP-023 monotherapy
  Interventions: Drug: IDP-023; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase 2: Combination IDP-023 plus rituximab (Experimental): NHL patients treated with multiple doses of IDP-023 in combination with rituximab
  Interventions: Drug: IDP-023; Drug: Rituximab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase 2: Combination IDP-023 plus daratumumab (Experimental): MM patients treated with multiple doses of IDP-023 in combination with daratumumab
  Interventions: Drug: IDP-023; Drug: Daratumumab; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna
- Phase 2: Combination IDP-023 plus isatuximab (Experimental): MM patients treated with multiple doses of IDP-023 in combination with isatuximab
  Interventions: Drug: IDP-023; Drug: Interleukin-2; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mesna; Drug: Isatuximab

INTERVENTIONS:
Drug: IDP-023 — NK cell therapy
Drug: Rituximab — Anti-CD20 antibody therapy
  Other Names: Rituxan
  Arms: Phase 2: Combination IDP-023 plus rituximab
Drug: Daratumumab — Anti-CD38 antibody therapy
  Other Names: Darzalex
  Arms: Phase 2: Combination IDP-023 plus daratumumab
Drug: Interleukin-2 — Immune cytokine
  Other Names: Proleukin
  Arms: Phase 1: Single Agent IDP-023 - Multiple Doses with IL-2; Phase 2: Combination IDP-023 plus daratumumab; Phase 2: Combination IDP-023 plus isatuximab; Phase 2: Combination IDP-023 plus rituximab
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy
Drug: Mesna — Chemoprotectant
Drug: Isatuximab — Anti-CD38 antibody therapy
  Other Names: Sarclisa
  Arms: Phase 2: Combination IDP-023 plus isatuximab

SUMMARY:
This is an open label, Phase 1/2, first-in-human, multiple ascending dose, and dose-expansion study of IDP-023 administered as a single agent and in combination with or without interleukin-2 (IL-2), and with or without isatuximab, daratumumab or rituximab to evaluate the safety, tolerability and preliminary antitumor activity in patients with advanced hematologic cancers.

DETAILED DESCRIPTION:
IDP-023 is an off-the-shelf, allogeneic cell product made of "natural killer" cells, also called NK cells. White blood cells are part of the immune system and NK cells are a type of white blood cell that are known to kill cancer cells.

This is an open label, Phase 1/2, first-in-human, multiple ascending dose, and dose-expansion study of IDP-023 administered as a single agent and in combination with or without interleukin-2 (IL-2), and with or without isatuximab, daratumumab or rituximab to evaluate the safety, tolerability, and preliminary antitumor activity in patients with relapsed and/or refractory advanced multiple myeloma (MM) or non-Hodgkin's lymphoma (NHL), respectively.

The study is divided into a phase 1 dose escalation phase and a phase 2 expansion phase.

Phase 1 (Escalation Phase): The primary objectives of Phase 1 are to define the safety of different IDP-023 containing regimens and to define the recommended regimen and Phase 2 doses (RP2D) of IDP-023.

Phase 2 (Expansion Phase): The objective of the Phase 2 expansion cohort is to evaluate the safety and efficacy of IDP-023 in advanced MM in combination with isatuximab or daratumumab and advanced NHL in combination with rituximab.

ELIGIBILITY:
Key Inclusion Criteria:

* For MM patients: Documented diagnosis of MM requiring systemic therapy and relapsed and/or refractory (R/R) disease after ≥ 3 prior lines of therapy.
* For NHL patients: R/R disease and failed ≥ 2 lines of systemic chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of greater than 12 weeks per the Investigator.

Key Exclusion Criteria:

* Impaired cardiac function or history of clinical significant cardiac disease.
* Human immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* Active SARS-CoV-2 infection.
* Has untreated central nervous system, epidural tumor metastasis, or brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Phase 1) | 1 year
  Escalation Period
Incidence of dose-limiting toxicities (DLTs) of IDP-023 Monotherapy - (Phase 1) | up to 21 days
  Escalation Period
Nature of dose-limiting toxicities (DLTs) of IDP-023 Monotherapy - (Phase 1) | up to 21 days
  Escalation Period
Incidence of dose-limiting toxicities (DLTs) of IDP-023 in combination with Isatuximab, Daratumumab or Rituximab - (Phase 1) | up to 35 days
  Escalation Period
Nature of dose-limiting toxicities (DLTs) of IDP-023 in combination with Isatuximab, Daratumumab or Rituximab - (Phase 1) | up to 35 days
  Escalation Period
Maximum tolerable dose (MTD) or a tolerated dose below MTD - (Phase 1) | 1 year
  Escalation Period
For MM: Anti-tumor activity by objective response rate (ORR), complete response (CR), stringent complete response (sCR), very good partial response (VGPR), and partial response (PR) - (Phase 2) | 2 years
  Expansion period
For NHL: Anti-tumor activity by objective response rate (ORR) - (Phase 2) | 2 years
  Expansion period

SECONDARY OUTCOMES:
PK (Cmax) of IDP-023 - (Phase 1/2) | 2 years
  Escalation and expansion periods
PK (AUC) of IDP-023 - (Phase 1/2) | 2 years
  Escalation and expansion periods
For MM: Anti-tumor activity by objective response rate (ORR), complete response (CR), stringent complete response (sCR), very good partial response (VGPR), and partial response (PR) - (Phase 1) | 1 year
  Escalation period
For NHL: Anti-tumor activity by objective response rate (ORR) - (Phase 1) | 1 year
  Escalation period
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Phase 2) | 2 years
  Expansion period

CONTACTS AND LOCATIONS:
Overall Officials: Indapta Therapeutics, Inc., Study Director — Indapta Therapeutics, INC.
Locations (12):
- United States (12):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Florida Cancer Specialists and Research Institute - Lake Mary Cancer Center, Lake Mary, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - NYP/Weill Cornell Medical Center, New York, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No